CLINICAL TRIAL: NCT04253691
Title: Sleep Intervention for Chronic Insomnia Using Virtual Reality Pilot Study
Acronym: iVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017122
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insomnia Chronic; Pain, Chronic
Keywords: Sleep; Pain; Virtual Reality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Virtual Reality Based Relaxation Therapy (Experimental): This is a pilot trial with one treatment condition (VR mediation).
  Interventions: Device: Virtual Reality Mediated Relaxation

INTERVENTIONS:
Device: Virtual Reality Mediated Relaxation — Participants will use a brief Virtual Reality relaxation protocol to improve their insomnia. Their workbook will contain a handout that outlines the details. Participants will be encouraged to refer to it at home if they forget any part of the procedure.

SUMMARY:
Sleep disturbances are common among chronic pain patients, with reports typically ranging from 50-70% of patients reporting sleep difficulties. It is well documented that, alongside a high comorbidity with chronic pain, chronic insomnia also has high comorbidity with, and is a risk factor for, developing an anxiety disorders. This clinical trial will examine the effects of virtual reality (VR) meditation environments on patients with pain- and insomnia-related anxiety. The purpose of this study is to examine the benefits of using VR meditation with patients with chronic pain and chronic sleep disturbance so that clinicians can more effectively treat core causes to symptoms and reduce counterproductive therapies.

Research objectives include:

1. To examine the clinical and health characteristics, including sleep, pain, fatigue, cognitive abilities, and cardiovascular health in patients with chronic pain.
2. To examine changes in the primary clinical outcomes, including chronic pain, complaints of poor sleep, and fatigue.
3. To examine changes in the secondary clinical outcomes, including mood, daytime functioning, cognitive functioning, and cardiovascular health.
4. To examine the mechanistic variables, including arousal (heart rate variability, HRV) and CS (thermal response).

DETAILED DESCRIPTION:
Sleep disturbances are common among chronic pain patients, with reports typically ranging from 50-70% of patients reporting sleep difficulties. It is well documented that, alongside a high comorbidity with chronic pain, chronic insomnia also has high comorbidity with, and is a risk factor for, developing an anxiety disorders. Research has shown that Cognitive Behavioral Therapies (CBT) are efficacious in treating patient with comorbid insomnia and chronic pain (e.g., improvements in sleep parameters, normal sleep efficiency, reductions in pain severity. CBT addresses a number of factors involved in the maintenance of patient sleep and health issues, and a key piece of CBT for insomnia and pain is the reduction of worrisome thoughts, or anxiety related to sleep and pain issues. A common evidence-based strategy used for reducing anxiety and worry is the practice of relaxation. The aim of this study is to investigate the benefits of replacing treatment as usual (TAU) relaxation practices, with Virtual Reality (VR) mediation environments within CBT treatment.

Virtual Reality Meditation for Anxiety

There are few studies in the literature demonstrating a relationship between Virtual Reality (VR) - a computer generated environment that presents the user with a realistic three-dimensional space - and reductions in anxious symptomology. However, the results of those studies are very encouraging. In a case study, Tarrant and Cope treated 4 firefighters who had anxiety and anxiety-based disorders with a Positivity VR Experience. 3 of 4 treated patients exhibited increased left gamma symmetry, associated with approach behavior and increased mood, and 3 of 4 patients showed increases in State-Cheerfulness and Positive Affect. Tarrant and colleagues also conducted a pilot study, where they treated 14 patients who had moderate or higher levels of generalized anxiety with a 5-minute Mindfulness in Nature experience. Patients in the VR meditation group showed both global and regional decreases in Beta activity (i.e., decrease in frequencies associated with qualitatively anxious states and decreased self-reported State Anxiety. Overall, these results seem promising, as they provide preliminary evidence supporting that VR interventions may be a useful and effective tool for the treatment of elevated anxiety symptoms.

In summary, this clinical trial will examine the effects of VR meditation environments on patients with pain- and insomnia-related anxiety. The proposed study design will yield important information about the efficacy of VR meditation practices. The purpose of this study is to examine the benefits of using VR meditation with patients with chronic pain and chronic sleep disturbance so that clinicians can more effectively treat core causes to symptoms and reduce counterproductive therapies.

Ultimately, this research targets two important public health concerns, namely insomnia and chronic pain. Insomnia in the context of chronic pain has been relatively understudied. Thus, the results of the present study will provide unique insights into sleep and chronic pain and will advance knowledge in the fields of both sleep and pain. Although the results of this study will be specific to chronic pain patients, they will have broader implications for other medical populations likely to suffer from chronic pain and insomnia (i.e., cancer patients, older adults). The information gained has the potential to make a significant contribution to behavioral healthcare practices for a wide variety of disorders, not just insomnia and pain. Thus, this research has implications not only for future sleep and pain research but also for other types of treatment-related research.

2. Objectives

1. To examine the clinical and health characteristics, including sleep, pain, fatigue, cognitive abilities, and cardiovascular health in patients with chronic pain.
2. To examine changes in the primary clinical outcomes, including chronic pain, complaints of poor sleep, and fatigue.
3. To examine changes in the secondary clinical outcomes, including mood, daytime functioning, cognitive functioning, and cardiovascular health.
4. To examine the mechanistic variables, including arousal (heart rate variability, HRV) and CS (thermal response).

ELIGIBILITY:
General inclusion criteria:

1. 18+ years,
2. able to read and understand English,
3. pain and insomnia complaints for 6+ months,
4. diagnosed with (4.1) insomnia based on the criteria below:

4.1) insomnia complaints for 6+ months that:

4.1a) occur despite adequate opportunity and circumstances for sleep, and

4.1b) consist of 1 or more of the following: difficulty falling asleep, staying asleep, waking up too early, nonrestorative sleep,

4.1c) daytime dysfunction (mood, cognitive, social, occupational) due to insomnia,

4.1d) screening ISI score ≥ 11

Exclusion criteria:

1. unable to provide informed consent,
2. unable to complete forms and implement treatment due to cognitive impairment (MMSE<26),
3. sleep disorder other than insomnia (i.e., sleep apnea [apnea/hypopnea index, AHI>15], Periodic Limb Movement Disorder-PLMD [myoclonus arousals per hour > 15]),
4. bipolar or seizure disorder (due to risk of sleep restriction treatment),
5. other major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychotic disorders),
6. severe untreated psychiatric comorbidity,
7. psychotropic or other medications (e.g., beta-blockers) that alter pain or sleep,
8. participation in any nonpharmacological treatment (including CBT) for pain, sleep, fatigue or mood outside the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Daily Electronic Sleep/Pain Diaries | 6 weeks
  Daily electronic dairies will record pain intensity and unpleasantness, sleep (latency, wake after onset, efficiency, quality), fatigue, sleep and pain medication consumption
Objective Daily Sleep Actiwatch-2 (Wake After Sleep Onset) | 6 weeks
  Objective wake after sleep onset
Objective Daily Sleep Actiwatch-2 (Sleep Onset Latency) | 6 weeks
  Objective sleep onset latency
Objective Daily Sleep Actiwatch-2 (Sleep Efficiency) | 6 weeks
  Objective sleep efficiency
Insomnia Severity Index | 6 weeks
  Insomnia severity measurement; min: 0 max:28; higher score means greater insomnia severity
Fatigue Severity Scale | 6 weeks
  Fatigue severity; min:10 max: 73; higher score means higher fatigue severity

SECONDARY OUTCOMES:
Patient centered outcomes questionnaire | 6 weeks
  The Patient Centered Outcomes questionnaire assesses four domains (pain, fatigue, emotional distress, and interference with daily activities) relevant to chronic pain populations on a numerical rating scale ranging from 0-10; min: 0 max:200; 200; A greater score equates a worse outcome
Computerized Cognitive Assessments -WCST | 6 weeks
  Determine level of cognitive functioning
Computerized Cognitive Assessments - Stroop Task | 6 weeks
  Determine level of cognitive functioning
Computerized Cognitive Assessments - Sternberg tasks | 6 weeks
  Determine level of cognitive functioning
List learning-Rey Auditory Learning Test modified for visual presentation | 6 weeks
  Immediate and delayed recall memory
Beck Depression Inventory Second Edition | 6 weeks
  Depressive symptom assessment; min: 0 max: 63; Higher score means higher severity of depression
State Trait Anxiety Inventory | 6 weeks
  Assessment of Anxiety symptoms; mix: 0 max:60; higher score means higher anxiety
Cognitive Failures Questionnaire | 6 weeks
  Self-reported failures in perception, memory, and motor function; min:0 max: 100; higher score means greater cognitive failure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Tarrant J, Viczko J, Cope H. Virtual Reality for Anxiety Reduction Demonstrated by Quantitative EEG: A Pilot Study. Front Psychol. 2018 Jul 24;9:1280. doi: 10.3389/fpsyg.2018.01280. eCollection 2018. PMID 30087642
- [Background] Thompson, M., & Thompson, L. (2007). Neurofeedback for stress management. Principles and practice of stress management, 3, 249-287.
- [Background] Tarrant, J., & Cope, H. (2018). Combining frontal gamma asymmetry neurofeedback with virtual reality: A proof-of-concept case study. NeuroRegulation, 5(2), 57-66. https://doi.org/10.15540/nr.5.2.57
- [Background] Sutton, S. K., & Davidson, R. J. (1997). Prefrontal Brain Asymmetry: A Biological Substrate of the Behavioral Approach and Inhibition Systems. Psychological Science, 8(3), 204-210. https://doi.org/10.1111/j.1467-9280.1997.tb00413.x
- [Background] Price, J., & Budzynski, T. (2009). Anxiety, EEG patterns, and neurofeedback. Introduction to quantitative EEG and neurofeedback: Advanced theory and applications, 453-470.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04253691/Prot_SAP_000.pdf